CLINICAL TRIAL: NCT05507515
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Five-part Study to Assess the Safety, Tolerability, and Pharmacokinetics of Single and Multiple Oral Doses of ONO-2020 in Healthy Participants
Brief Title: A Phase 1 Study of ONO-2020 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ONO-2020-01
Record Dates: First submitted 2022-08-11; First posted 2022-08-19 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (16):
- Part A: Cohort A1 ONO-2020 or Placebo - fasted (Experimental): Single ascending doses of ONO-2020 orally under fasted conditions
  Interventions: Drug: ONO-2020; Drug: Placebo
- Part A: Cohort A2 ONO-2020 or Placebo - fasted and fed (Experimental): Single ascending doses of ONO-2020 orally under fasted and fed conditions
  Interventions: Drug: ONO-2020; Drug: Placebo
- Part A: Cohort A3 ONO-2020 or Placebo - fasted (Experimental): Single ascending doses of ONO-2020 orally under fasted conditions
  Interventions: Drug: ONO-2020; Drug: Placebo
- Part A: Cohort A4 ONO-2020 or Placebo - fasted and fed (Experimental): Single ascending doses of ONO-2020 orally under fasted and fed conditions
  Interventions: Drug: ONO-2020; Drug: Placebo
- Part A: Cohort A5 ONO-2020 or Placebo - fasted (Experimental): Single ascending doses of ONO-2020 orally under fasted conditions
  Interventions: Drug: ONO-2020; Drug: Placebo
- Part A: Cohort A6 ONO-2020 or Placebo - fasted (Experimental): Single ascending doses of ONO-2020 orally under fasted conditions
  Interventions: Drug: ONO-2020; Drug: Placebo
- Part B: Cohort B1 ONO-2020 or Placebo (Experimental): Multiple ascending doses of ONO-2020 orally for 14 days
  Interventions: Drug: ONO-2020; Drug: Placebo
- Part B: Cohort B2 ONO-2020 or Placebo (Experimental): Multiple ascending doses of ONO-2020 orally for 14 days
  Interventions: Drug: ONO-2020; Drug: Placebo
- Part B: Cohort B3 ONO-2020 or Placebo (Experimental): Multiple ascending doses of ONO-2020 orally for 14 days
  Interventions: Drug: ONO-2020; Drug: Placebo
- Part B: Cohort B4 ONO-2020 or Placebo (Experimental): Multiple ascending doses of ONO-2020 orally for 14 days
  Interventions: Drug: ONO-2020; Drug: Placebo
- Part B: Cohort B5 ONO-2020 or Placebo (Experimental): Multiple ascending doses of ONO-2020 orally for 14 days
  Interventions: Drug: ONO-2020; Drug: Placebo
- Part C: Cohort C1 ONO-2020 (Experimental): Single dose of ONO-2020 orally for CSF sampling
  Interventions: Drug: ONO-2020
- Part C: Cohort C2 ONO-2020 (Experimental): Single dose of ONO-2020 orally for CSF sampling
  Interventions: Drug: ONO-2020
- Part D: Cohort D1 ONO-2020 or Placebo (Experimental): Single dose of ONO-2020 orally in elderly healthy volunteers
  Interventions: Drug: ONO-2020; Drug: Placebo
- Part E: Cohort E1 ONO-2020 or Placebo (Experimental): Multiple ascending doses of ONO-2020 orally for 14 days in Japanese healthy volunteers
  Interventions: Drug: ONO-2020; Drug: Placebo
- Part E: Cohort E2 ONO-2020 or Placebo (Experimental): Multiple ascending doses of ONO-2020 orally for 14 days in Japanese healthy volunteers
  Interventions: Drug: ONO-2020; Drug: Placebo

INTERVENTIONS:
Drug: ONO-2020 — ONO-2020 tablets
Drug: Placebo — Placebo tablets matching ONO-2020 tablets
  Arms: Part A: Cohort A1 ONO-2020 or Placebo - fasted; Part A: Cohort A2 ONO-2020 or Placebo - fasted and fed; Part A: Cohort A3 ONO-2020 or Placebo - fasted; Part A: Cohort A4 ONO-2020 or Placebo - fasted and fed; Part A: Cohort A5 ONO-2020 or Placebo - fasted; Part A: Cohort A6 ONO-2020 or Placebo - fasted; Part B: Cohort B1 ONO-2020 or Placebo; Part B: Cohort B2 ONO-2020 or Placebo; Part B: Cohort B3 ONO-2020 or Placebo; Part B: Cohort B4 ONO-2020 or Placebo; Part B: Cohort B5 ONO-2020 or Placebo; Part D: Cohort D1 ONO-2020 or Placebo; Part E: Cohort E1 ONO-2020 or Placebo; Part E: Cohort E2 ONO-2020 or Placebo

SUMMARY:
The purpose of this FIH study is to evaluate the safety, tolerability and pharmacokinetics of ONO-2020 in healthy adult participants. This FIH study consists of five parts (Parts A-E) to study single or multiple doses of ONO-2020 in healthy participants, including elderly and Japanese participants, as well as the food effect on the PK of ONO-2020. These data will support the clinical development program and help inform dose selection in future studies.

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 55 years of age (Parts A, B, C, and E) or ≥65 years of age (Part D) inclusive at the time of informed consent.
2. Male and female participants of non-Japanese ethnicity (Parts A, B, C, and D) or of Japanese ethnicity (Part E).
3. No clinically significant medical history and no abnormal physical examination, laboratory profiles, vital signs or ECG abnormalities, based on the Screening examination.
4. Body mass index of ≥18.5 to <30 kg/m2, and a body weight of at least 50 kg for males and 45 kg for females to a maximum of 100 kg, at the time of Screening.
5. Agree to use an effective method of contraception.
6. Able and willing to give informed consent after reading the information and consent form and after having the opportunity to discuss the study with the Investigator or designee.
7. Estimated creatinine clearance (CrCL, Cockcroft-Gault equation) ≥90 mL/min at Screening. In Part D only, an estimated ≥60 mL/min at Screening.
8. Fully vaccinated for SARS-CoV-2 (received primary series of COVID-19 vaccine) prior to Screening.

Exclusion Criteria:

1. Mentally or legally incapacitated or has significant emotional problems at the time of the Screening visit or expected during the conduct of the study.
2. History or presence of clinically significant medical, surgical or psychiatric condition or disease that in the opinion of the Investigator or Sponsor Medical Monitor might confound the results of the study or pose an additional risk to the participant by their participation in the study.
3. hypersensitivity or idiosyncratic reaction to the study interventions, excipients or related compounds, or severe food allergies.
4. alcoholism or drug/chemical/substance abuse within the past 2 years prior to the first dosing.
5. Use of any drug, including prescription and non-prescription medications, herbal remedies, or vitamin supplements, including St. John's Wort, within 14 days or five half-lives (whichever is longer) of first dosing and throughout the study.
6. Use of any drugs known to be significant inducers or inhibitors of cytochrome P450 (CYP) enzymes and/or drug transporter substrates for 28 days prior to the first dosing and throughout the study.
7. Participation in another clinical study within 120 days (or five half-lives of the study intervention, whichever is longer) prior to the first dosing.
8. Liver function test values are in the abnormal range before inclusion.
9. Positive urine drug, alcohol, or cotinine results at Screening or check in.
10. Positive results at Screening for active viral infection that include HIV, HBV, HCV, and SARS-CoV-2.
11. Seated resting blood pressure is less than 90/40 mmHg or greater than 140/90 mmHg at Screening.
12. Seated resting pulse rate is lower than 40 beats per minute (bpm) or higher than 100 bpm at Screening.
13. Clinically significant history or presence of ECG findings.
14. The participant is a current smoker or has smoked within 3 months of Screening or has a positive urine cotinine at Screening or admission.
15. Female who is pregnant or lactating.
16. Donation of blood or significant blood loss of 400 mL or more within 90 days prior to the first dosing, or blood donation of 200 mL or more within 30 days prior to the first dosing, or blood plasma or platelet donation within 14 days prior to the first dosing, or blood transfusion within 90 days prior to the first dosing.
17. Participants who, in the opinion of the Investigator, are considered unsuitable for any other reason.

    Exclusion criteria, applicable to all participants taking part in the food effect Cohort in Part A:
18. Participants who are vegetarian or vegan or not willing to eat a high-fat breakfast.

    Exclusion criteria, applicable to all participants undergoing lumbar puncture for CSF collection (Part C):
19. History of significant back pain, significant kyphosis, and or scoliosis or other spinal column deformities.
20. History of poor venous access.
21. History of hypersensitivity for local anesthetics (Lidocaine).
22. History or evidence or fundoscopic findings suggestive of raised intracranial pressure.
23. History or evidence of laboratory abnormalities for coagulation parameters or the use of medications that may increase the risk of bleeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2022-07-29 (Actual); Primary Completion 2023-12-24 (Actual); Study Completion 2023-12-24 (Actual)

PRIMARY OUTCOMES:
Incidence, severity, and type of treatment emergent adverse events (TEAEs) | Part A, C and D: From screening up to Day 7, Part B and E: From screening up to Day 21
  Incidence of TEAEs will be summarized overall, and by study part and dose group using frequency and percentage.
Vital signs (blood pressure) | Part A, C and D: From screening up to Day 7, Part B and E: From screening up to Day 21
  Observed values and change from baseline results will be summarized by analysis time point, and summaries of clinically significant and non-clinically significant abnormalities will be provided by each time point.
Vital signs (pulse rate) | Part A, C and D: From screening up to Day 7, Part B and E: From screening up to Day 21
  Observed values and change from baseline results will be summarized by analysis time point, and summaries of clinically significant and non-clinically significant abnormalities will be provided by each time point.
Vital signs (body temperature) | Part A, C and D: From screening up to Day 7, Part B and E: From screening up to Day 21
  Observed values and change from baseline results will be summarized by analysis time point, and summaries of clinically significant and non-clinically significant abnormalities will be provided by each time point.
Vital signs (respiratory rate) | Part A, C and D: From screening up to Day 7, Part B and E: From screening up to Day 21
  Observed values and change from baseline results will be summarized by analysis time point, and summaries of clinically significant and non-clinically significant abnormalities will be provided by each time point.
12-lead electrocardiograms (ECGs) parameters, such as but not limited to heart rate, RR, PR, QRS, QT, and corrected QT intervals (QTcF) | Part A, C and D: From screening up to Day 7, Part B and E: From screening up to Day 21
  The number and percentage of subjects with normal, abnormal not clinically significant and abnormal clinically significant of ECG results will be tabulated at each time point.
Clinically significant abnormal telemetry electrocardiograms (ECGs) | Part A and D: Day 1
  The number and percentage of subjects with normal, abnormal not clinically significant and abnormal clinically significant of telemetry ECGs results will be tabulated at each time point.
Clinically significant abnormal physical examination findings | Part A, C and D: From screening up to Day 7, Part B and E: From screening up to Day 21
  The number and percentage of subjects with normal, abnormal not clinically significant and abnormal clinically significant of physical examination results will be tabulated at each time point.
Clinical laboratory abnormalities (hematology, clinical chemistry, coagulation, and urinalysis) | Part A, C and D: From screening up to Day 7, Part B and E: From screening up to Day 21
  The number and percentage of subjects with abnormal laboratory results at any time during the study will be tabulated.
Ophthalmologic examination findings (pupil size and pupillary light reflex) | Part A, C and D: From Day 1 up to Day 7, Part B and E: From Day 1 up to Day 21
  The number and percentage of subjects with miosis will be summarized by laterality at each time point.
Clinically abnormal findings in Mini-International Neuropsychiatric Interview Screen (M.I.N.I.-Screen) | Part A, C and D: From screening up to Day 7, Part B and E: From screening up to Day 21
  Responses to the M.I.N.I.-Screen will be listed.
Clinically abnormal findings in Columbia Suicide Severity Rating Scale (C-SSRS) | Part A, C and D: From screening up to Day 7, Part B and E: From screening up to Day 21
  Responses to the suicidality assessment scale (C-SSRS) will be listed.

SECONDARY OUTCOMES:
Pharmacokinetics (Cmax in plasma) | Part A, C and D: Day 1 through Day 4, Part B and E: Day 1 through Day 19
Pharmacokinetics (Tmax in plasma) | Part A, C and D: Day 1 through Day 4, Part B and E: Day 1 through Day 19
Pharmacokinetics (AUClast in plasma) | Part A, C and D: Day 1 through Day 4, Part B and E: Day 1 through Day 19
Pharmacokinetics (AUCinf in plasma) | Part A, C and D: Day 1 through Day 4, Part B and E: Day 1 through Day 19
Pharmacokinetics (T1/2 in plasma) | Part A, C and D: Day 1 through Day 4, Part B and E: Day 1 through Day 19
Pharmacokinetics (CL/F in plasma) | Part A, C and D: Day 1 through Day 4, Part B and E: Day 1 through Day 19
Pharmacokinetics (Aet in urine) | Part A and D: Day 1 through Day 4
Pharmacokinetics (fe/F in urine) | Part A and D: Day 1 through Day 4
Pharmacokinetics (CLR in urine) | Part A and D: Day 1 through Day 4
Pharmacokinetics (Ctrough in plasma) | Part B and E: Day 2 through Day 13
Pharmacokinetics (ONO-2020 concentration in CSF) | Part C: Day 2

CONTACTS AND LOCATIONS:
Overall Officials: Project Leader, Study Director — Ono Pharma USA Inc
Locations (1):
- Altasciences, Cypress, California, United States

IPD SHARING:
Plan to Share IPD: No